CLINICAL TRIAL: NCT04953182
Title: Around the Clock Pain Treatment Modality Offer Better Pain Control and Less Opiates Drugs Use
Brief Title: Pain Modality Treatment After Hemorrhoidectomy
Status: Completed | Type: Observational
Sponsor: Assuta Medical Center (Other)
Responsible Party: Principal Investigator, Sergio Gabriel Susmallian, Head of the department of general surgery, Assuta Medical Center
Other Study IDs: 12-2020
Record Dates: First submitted 2021-06-26; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Pain, Acute; Pain, Procedural
Keywords: Pain killers
MeSH Terms: conditions — Acute Pain; Pain, Procedural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Around the clock analgetic treatment: Patients that underwent hemorrhoidectomy and pain killers are prescribed every specific hour independent of pain degree, if necessary drugs can be administered on demand.
  Interventions: Other: Pain scale registry
- On demand analgetic treatment: A pain killers list is prescribed by the physician and the nurse decides which drug to administer depending on a protocol of treatment based on the visual analog scale.
  Interventions: Other: Pain scale registry

INTERVENTIONS:
Other: Pain scale registry — The nurses ask the patient about the pain filling every two hours during the hospitalization.

SUMMARY:
Hemorrhoidectomy is one of the operations that causes the greatest intensity of pain. Treatment of postoperative pain is essential for the well-being of the patient. Long-term use of opioids and different drugs can have unintended consequences.

The objective is to corroborate which pain treatment modality is better in patients after hemorrhoidectomy.

DETAILED DESCRIPTION:
Patients who have undergone a hemorrhoidectomy are included in the study, the pain treatment modality is conceived by the treating surgeon or anesthesiologist. The first modality is to administer pain killers on-demand depending on visual analog scales of pain and the second modality to give pain killers on determined hours.

ELIGIBILITY:
Inclusion Criteria:

Elective surgery for hemorrhoids

Exclusion Criteria:

Mental retardation Incapacitated patient Under 18 years old

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients that underwent elective hemorrhoidectomy
Sampling Method: Non-Probability Sample
Enrollment: 5335 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Pain medition | Immediately after the intervention/procedure/surgery
  The pain registred is analyze as maximum, mean and on discharge.
Drugs Administred | Immediately after the intervention/procedure/surgery
  The amount of drugs administred to each patients is analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Sergio G Susmallian, MD, Principal Investigator — Assuta Medical Center

IPD SHARING:
Plan to Share IPD: No
The data will be sent to the accepting journal study

REFERENCES:
- [Derived] Susmallian S, Aviv I, Babis I, Segal E. Analysis of Two Treatment Modalities for Post-surgical Pain after Hemorrhoidectomy. Chirurgia (Bucur). 2024 Jun;119(3):247-259. doi: 10.21614/chirurgia.2024.v.119.i.3.p.247. PMID 38982903